CLINICAL TRIAL: NCT01745172
Title: Carotid Body Removal for the Treatment of Chronic Diseases Characterized by Excessive Central Sympathetic Activity Including Resistant Hypertension: a Pilot Study.
Brief Title: Carotid Body Removal for the Treatment of Resistant Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noblewell (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBR-BRISTOL.UK-CIBIEM
Record Dates: First submitted 2012-11-22; First posted 2012-12-10 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carotid body excision (Experimental): Patients undergoing the carotid body excision to test the hypothesis that carotid body excision is sufficient to attain target blood pressure.
  Interventions: Procedure: Carotid body excision

INTERVENTIONS:
Procedure: Carotid body excision — This surgery does not involve any study drug or investigational device.
  The carotid body will be removed by the so called 'lateral approach' or a combined 'lateral and medial approach'. In all cases the target area was defined as the tissue in between the ECA and ICA, up to 5-6mm above the bifurcation point of the common carotid artery into the ECA and ICA. In a lateral approach the carotid bifurcation is not turned. A combined approach includes usually dissection of the superior thyroid vessel and turning of the carotid bifurcation.

SUMMARY:
This is a pilot study to assess the effectiveness, safety and feasibility of carotid body removal in patients with high blood pressure (hypertension) resistant to medical treatment. Patients with high blood pressure are at significant risk of medical complications including stroke and heart disease. The principle research question is whether removal of the carotid body will lead to an improvement in the blood pressure of this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Age of participants will be 18-75 years
* Resistant HTN criteria:

  1. Daytime mean ambulatory systolic blood pressure ≥135mmHg and office systolic blood pressure ≥150mmHg
  2. Patients on at least three anti-hypertensive medications, including a diuretic, at maximum tolerated dose
  3. No evidence of causes for secondary HTN following thorough clinical assessment
  4. Patient medication concordance will be monitored via medication/blood pressure diary

Exclusion Criteria:

* Calculated GFR <45ml/min/1.73m2
* Carotid body located outside the defined carotid septum
* Obstructive carotid atherosclerotic disease with >50% stenosis
* Oxygen desaturation at rest below 92%
* Known structural lung disease
* Requirement for oxygen therapy to maintain oxygen saturation
* Patients wish to participate in mountain climbing, skin diving or free diving
* Pregnancy or anticipation of pregnancy
* Palliative care/chemotherapy
* Acute coronary syndrome or unstable angina
* Stroke or transient ischaemic attack (TIA) < 6 months prior to procedure
* Expected life expectancy less than 12 months due to other disease
* Intravenous drug use
* Alcohol intake >28 units/week
* Febrile illness within two weeks of participation
* Unable to attend for follow up appointments in Bristol at 1, 3, 6, 12 and 24 months post-operatively.

MR imaging related exclusion criteria (all participants):

* Pace-maker, implantable cardiac defibrillator, cerebral metallic clips or other implanted metal devices/structures
* Unable to tolerate scanner or history of panic attacks/claustrophobia
* Learning disability, significant hearing or visual impairment (participant would need to able to communicate from within the MRI scanner)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change of Blood Pressure | Baseline and 3 months
  Change from Baseline Blood Pressure at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Sobotka, MD, Study Director — Cibiem, Inc.
Locations (1):
- Clinical Research and Imaging Centre (CRIC) and the Bristol Heart Institute (BHI), University Hospitals Bristol NHS Foundation Trust, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes